CLINICAL TRIAL: NCT01120028
Title: Open-label, Randomised Multicentre Study of CAMPATH-1H Versus Basiliximab Induction Treatment and Sirolimus Versus Tacrolimus Maintenance Treatment for the Preservation of Renal Function in Patients Receiving Kidney Transplants
Brief Title: Campath, Calcineurin Inhibitor Reduction and Chronic Allograft Nephropathy
Acronym: 3C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Health Service, United Kingdom (Other Government); Pfizer (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CTSU3C1; 2008-008553-27 (EudraCT Number); ISRCTN88894088 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Alemtuzumab; Sirolimus; Basiliximab; Tacrolimus; Campath-1H
MeSH Terms: interventions — Alemtuzumab; Basiliximab; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Alemtuzumab/Sirolimus (Experimental): Induction therapy allocation: Alemtuzumab (Campath-1H).
  Maintenance therapy allocation (at 6-months post-transplant): Sirolimus
  Interventions: Drug: Alemtuzumab; Drug: Sirolimus
- Alemtuzumab/Tacrolimus (Experimental): Induction therapy allocation: Alemtuzumab (Campath-1H).
  Maintenance therapy allocation (at 6-months post-transplant): Tacrolimus
  Interventions: Drug: Alemtuzumab; Drug: Tacrolimus
- Basiliximab/Tacrolimus (Active Comparator): Induction therapy allocation: Basiliximab.
  Maintenance therapy allocation (at 6-months post-transplant): Tacrolimus
  Interventions: Drug: Basiliximab; Drug: Tacrolimus
- Basiliximab/Sirolimus (Active Comparator): Induction therapy allocation: Basiliximab.
  Maintenance therapy allocation (at 6-months post-transplant): Sirolimus
  Interventions: Drug: Basiliximab; Drug: Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab 30 mg intravenously or subcutaneously, two doses 24 hours apart
  Other Names: Campath-1H
  Arms: Alemtuzumab/Sirolimus; Alemtuzumab/Tacrolimus
Drug: Basiliximab — 20 mg intravenously, two doses 96 hours apart
  Other Names: Simulect
  Arms: Basiliximab/Sirolimus; Basiliximab/Tacrolimus
Drug: Sirolimus — Sirolimus: target trough levels 6-12 ng/mL for first 6-months after maintenance therapy randomization, then 5-10 ng/mL
  Other Names: Rapamune
  Arms: Alemtuzumab/Sirolimus; Basiliximab/Sirolimus
Drug: Tacrolimus — Tacrolimus: target trough levels 5-7 ng/mL after maintenance therapy randomization.
  Other Names: Prograf
  Arms: Alemtuzumab/Tacrolimus; Basiliximab/Tacrolimus

SUMMARY:
The 3C study is investigating whether reducing exposure to calcineurin inhibitors (by using more potent antibody induction treatment and/or an elective switch to sirolimus) can improve the function and survival of kidney transplants.

DETAILED DESCRIPTION:
The long-term survival of kidney transplants has not improved over the past decade despite reductions in the rate of acute rejection. The commonest cause of late graft loss is chronic allograft nephropathy which is frequently caused by calcineurin inhibitor toxicity. Therefore, it may be possible to improve long-term graft outcomes by reducing the amount of calcineurin inhibitor exposure.

Two possible strategies to do this were tested. Firstly, Campath-1H (a monoclonal lymphocyte-depleting antibody) was compared to standard basiliximab-based induction. All patients then received tacrolimus-based maintenance therapy for 6-months (using lower doses in the Campath-1H arm).

At six months, patients were re-randomized between remaining on tacrolimus and converting to sirolimus (and therefore no longer taking calcineurin inhibitors). Patients were then followed-up in clinic and through routine NHS registries to collect information on relevant outcomes (including graft function, survival, hospitalisations and death).

ELIGIBILITY:
Inclusion Criteria:

* men or women aged over 18 years
* recipient of kidney transplant (planned in next 24 hours)

Exclusion Criteria:

* recipients of multi-organ transplant
* previous treatment with Campath-1H
* active infection (including HIV, hepatitis B or C)
* history of anaphylaxis to humanized monoclonal antibody
* history of malignancy (except adequately treated non-melanoma skin cancer)
* loss of kidney transplant within 6 months not due to technical reasons
* medical history that might limit the individual's ability to take trial treatments for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Friend, Study Director — University of Oxford; Colin Baigent, Principal Investigator — University of Oxford; Martin J Landray, Principal Investigator — University of Oxford; Paul Harden, Principal Investigator — University of Oxford; Richard Haynes, Principal Investigator — University of Oxford
Locations (20):
- United Kingdom (20):
  - Oxford Radcliffe Hospitals NHS Trust, Oxford, Oxon
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital NHS Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - University Hospitals Coventry & Warwickshire, Coventry
  - Royal Infirmary, Edinburgh
  - Western Infirmary, Glasgow
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Bart's and the London NHS Trust, London
  - Guy's and St Thomas's NHS Trust, London
  - Kings College Hospital NHS Trust, London
  - Royal Free Hampstead NHS Trust, London
  - Central Manchester NHS Trust, Manchester
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Plymouth Teaching Hospitals NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Sheffield Teaching Hospitals NHS Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Proposals for substudies must be approved by the Steering Committee. Procedure for accessing the data for this study are available on https://www.ndph.ox.ac.uk/data-access
Supporting Information: Study Protocol, SAP
Access Criteria: See URL
URL: https://www.ndph.ox.ac.uk/data-access

REFERENCES:
- [Result] 3C Study Collaborative Group; Haynes R, Harden P, Judge P, Blackwell L, Emberson J, Landray MJ, Baigent C, Friend PJ. Alemtuzumab-based induction treatment versus basiliximab-based induction treatment in kidney transplantation (the 3C Study): a randomised trial. Lancet. 2014 Nov 8;384(9955):1684-90. doi: 10.1016/S0140-6736(14)61095-3. Epub 2014 Jul 28. PMID 25078310
- [Result] 3C Study Collaborative Group. Campath, calcineurin inhibitor reduction, and chronic allograft nephropathy (the 3C Study) - results of a randomized controlled clinical trial. Am J Transplant. 2018 Jun;18(6):1424-1434. doi: 10.1111/ajt.14619. Epub 2018 Jan 9. PMID 29226570
- [Derived] Haynes R, Baigent C, Harden P, Landray M, Akyol M, Asderakis A, Baxter A, Bhandari S, Chowdhury P, Clancy M, Emberson J, Gibbs P, Hammad A, Herrington W, Jayne K, Jones G, Krishnan N, Lay M, Lewis D, Macdougall I, Nathan C, Neuberger J, Newstead C, Pararajasingam R, Puliatti C, Rigg K, Rowe P, Sharif A, Sheerin N, Sinha S, Watson C, Friend P; 3C Study Collaborative Group. Campath, calcineurin inhibitor reduction and chronic allograft nephropathy (3C) study: background, rationale, and study protocol. Transplant Res. 2013 May 6;2(1):7. doi: 10.1186/2047-1440-2-7. PMID 23641902
- See also: 3C study website — http://www.3cstudy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3C was conducted in 18 transplant centres in the UK. Recruitment took place between October 2010 and July 2013.
Pre-assignment Details: 852 participants were randomized for a comparison of Alemtuzumab (426) and Basiliximab (426) based induction therapies. After 6-months, 394 of those participants were re-randomized to either Sirolimus (197) or Tacrolimus (197) based maintenance therapies.
Groups:
- Period 1: Alemtuzumab/Tacrolimus: Induction therapy allocation: Alemtuzumab (Campath-1H) and Tacrolimus
  Alemtuzumab: Alemtuzumab 30 mg intravenously or subcutaneously, two doses 24 hours apart
  Tacrolimus: Target trough level 5-7 ng/mL for 6-months after alemtuzumab.
- Period 1: Basiliximab/Tacrolimus: Induction therapy allocation: Basiliximab and Tacrolimus
  Basiliximab: 20 mg intravenously, two doses 96 hours apart
  Tacrolimus: Target trough level 5-12 ng/mL for 6-months after basiliximab
- Period 2: Sirolimus: Sirolimus maintenance therapy: target trough level of 6-12 ng/mL for the first 6-months, then reducing to 5-10 ng/mL.
- Period 2: Tacrolimus: Tacrolimus maintenance therapy: target trough level of 5-7 ng/mL
Period: Period 1: Alemtuzumab or Basiliximab
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus | Period 2: Sirolimus | Period 2: Tacrolimus
Started | 426 | 426 | 0 | 0
Completed | 412 | 403 | 0 | 0
Not Completed | 14 | 23 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 0
Not completed — Not transplanted | 14 | 18 | 0 | 0
Period: Period 2: Tacrolimus or Sirolimus
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus | Period 2: Sirolimus | Period 2: Tacrolimus
Started | 0 | 0 | 197 | 197
Completed | 0 | 0 | 197 | 197
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
Groups:
- Period 1: Alemtuzumab/Tacrolimus: Induction therapy allocation: Alemtuzumab (Campath-1H) and Tacrolimus
  Alemtuzumab: Alemtuzumab 30 mg intravenously or subcutaneously, two doses 24 hours apart.
  Tacrolimus: Target trough level 5-7 ng/mL for 6-months after alemtuzumab.
- Period 1: Basiliximab/Tacrolimus: Induction therapy allocation: Basiliximab and Tacrolimus
  Basiliximab: 20 mg intravenously, two doses 96 hours apart.
  Tacrolimus: Target trough level 5-12 ng/mL for 6-months after basiliximab.
- Total: Total of all reporting groups
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus | Period 2: Sirolimus | Period 2: Tacrolimus | Total
Number analyzed (Participants) | 426 | 426 | 197 | 197 | 1246
Age, Categorical [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Age, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Age, Period 1: <=18 years | 0 | 0 | 0 | 0 | 0
    Age, Period 1: Between 18 and 65 years | 347 | 350 | 0 | 0 | 697
    Age, Period 1: >=65 years | 79 | 76 | 0 | 0 | 155
    Age, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Age, Period 2: <=18 years | 0 | 0 | 0 | 0 | 0
    Age, Period 2: Between 18 and 65 years | 0 | 0 | 163 | 162 | 325
    Age, Period 2: >=65 years | 0 | 0 | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  years
    Age, Continuous, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Age, Continuous, Period 1 | 52.1 (13.3) | 51.8 (13.3) |  |  | 51.9 (13.3)
    Age, Continuous, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Age, Continuous, Period 2 |  |  | 51.7 (13.0) | 52.0 (12.9) | 51.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Sex, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Sex, Period 1: Female | 149 | 151 | 0 | 0 | 300
    Sex, Period 1: Male | 277 | 275 | 0 | 0 | 552
    Sex, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Sex, Period 2: Female | 0 | 0 | 65 | 65 | 130
    Sex, Period 2: Male | 0 | 0 | 132 | 132 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Ethnic origin, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Ethnic origin, Period 1: White | 370 | 372 | 0 | 0 | 742
    Ethnic origin, Period 1: Black | 21 | 21 | 0 | 0 | 42
    Ethnic origin, Period 1: Asian | 30 | 23 | 0 | 0 | 53
    Ethnic origin, Period 1: Other | 5 | 10 | 0 | 0 | 15
    Ethnic origin, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Ethnic origin, Period 2: White | 0 | 0 | 174 | 173 | 347
    Ethnic origin, Period 2: Black | 0 | 0 | 5 | 7 | 12
    Ethnic origin, Period 2: Asian | 0 | 0 | 13 | 15 | 28
    Ethnic origin, Period 2: Other | 0 | 0 | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants] — All 852 participants were recruited in the UK. Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    United Kingdom: Period 1: United Kingdom | 426 | 426 | 0 | 0 | 852
    United Kingdom: Period 2: United Kingdom | 0 | 0 | 197 | 197 | 394
Primary Renal Disease [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Primary Renal Disease: Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Primary Renal Disease: Period 1: Diabetic kidney disease | 51 | 49 | 0 | 0 | 100
    Primary Renal Disease: Period 1: Glomerulonephritis | 92 | 89 | 0 | 0 | 181
    Primary Renal Disease: Period 1: Polycystic kidney disease | 68 | 73 | 0 | 0 | 141
    Primary Renal Disease: Period 1: Chronic pyelonephritis | 23 | 16 | 0 | 0 | 39
    Primary Renal Disease: Period 1: Hypertension | 42 | 42 | 0 | 0 | 84
    Primary Renal Disease: Period 1: Renovascular disease | 7 | 6 | 0 | 0 | 13
    Primary Renal Disease: Period 1: Other | 143 | 151 | 0 | 0 | 294
    Primary renal disease, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Primary renal disease, Period 2: Diabetic kidney disease | 0 | 0 | 15 | 21 | 36
    Primary renal disease, Period 2: Glomerulonephritis | 0 | 0 | 50 | 40 | 90
    Primary renal disease, Period 2: Polycystic kidney disease | 0 | 0 | 47 | 34 | 81
    Primary renal disease, Period 2: Chronic pyelonephritis | 0 | 0 | 5 | 9 | 14
    Primary renal disease, Period 2: Hypertension | 0 | 0 | 14 | 24 | 38
    Primary renal disease, Period 2: Renovascular disease | 0 | 0 | 3 | 4 | 7
    Primary renal disease, Period 2: Other | 0 | 0 | 63 | 65 | 128
Other Previous Disease [Number; unit: participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  participants
    Diabetes: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Diabetes | 74 | 67 |  |  | 141
    Vascular Disease: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Vascular Disease | 57 | 49 |  |  | 106
    Cancer: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Cancer | 18 | 5 |  |  | 23
Previous renal replacement [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Haemodialysis | 243 | 214 | 0 | 0 | 457
    Peritoneal dialysis | 104 | 106 | 0 | 0 | 210
    Transplant | 3 | 3 | 0 | 0 | 6
    None | 76 | 103 | 0 | 0 | 179
HLA mismatch level [Count of Participants; unit: Participants] — HLA = human leucocyte antigen.
  Level 1: 0-0-0; Level 2: 0 HLA-DR and 0/1 HLA-B mismatches; Level 3: (0 HLA-DR and 2 HLA-B) or (1 HLA-DR and 0/1 HLA-B); Level 4: (1 HLA-DR and 2 HLA-B) or (2 HLA-DR).
  Level 1 being most favourable, Level 4 being least favourable. Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    HLA mismatch level, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    HLA mismatch level, Period 1: Level 1 | 45 | 47 | 0 | 0 | 92
    HLA mismatch level, Period 1: Level 2 | 94 | 94 | 0 | 0 | 188
    HLA mismatch level, Period 1: Level 3 | 196 | 193 | 0 | 0 | 389
    HLA mismatch level, Period 1: Level 4 | 91 | 92 | 0 | 0 | 183
    HLA mismatch level, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    HLA mismatch level, Period 2: Level 1 | 0 | 0 | 23 | 22 | 45
    HLA mismatch level, Period 2: Level 2 | 0 | 0 | 42 | 42 | 84
    HLA mismatch level, Period 2: Level 3 | 0 | 0 | 89 | 90 | 179
    HLA mismatch level, Period 2: Level 4 | 0 | 0 | 43 | 43 | 86
Previous transplant [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Previous transplant, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Previous transplant, Period 1: None | 390 | 392 | 0 | 0 | 782
    Previous transplant, Period 1: ≥1 | 36 | 34 | 0 | 0 | 70
    Previous transplant, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Previous transplant, Period 2: None | 0 | 0 | 181 | 181 | 362
    Previous transplant, Period 2: ≥1 | 0 | 0 | 16 | 16 | 32
Highly sensitised [Count of Participants; unit: Participants] — Highly sensitised is defined as calculated reaction frequency >85% where the calculated reaction frequency is the proportion of the general UK population that the participant is predicted to be sensitised against. Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Highly sensitized, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Highly sensitized, Period 1: Yes | 16 | 15 | 0 | 0 | 31
    Highly sensitized, Period 1: No | 410 | 411 | 0 | 0 | 821
    Highly sensitized, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Highly sensitized, Period 2: Yes | 0 | 0 | 4 | 7 | 11
    Highly sensitized, Period 2: No | 0 | 0 | 193 | 190 | 383
Virology serology [Number; unit: Participants] — CMV=cytomegalovirus; EBV=Epstein-Barr virus. Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    CMV-positive donor to negative recipient: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    CMV-positive donor to negative recipient | 104 | 102 |  |  | 206
    EBV-positive donor to negative recipient: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    EBV-positive donor to negative recipient | 21 | 19 |  |  | 40
Type of donor [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    Type of donor, Period 1: number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Type of donor, Period 1: Donation after brain death | 148 | 145 | 0 | 0 | 293
    Type of donor, Period 1: Donation after circulatory death | 158 | 158 | 0 | 0 | 316
    Type of donor, Period 1: Donation from living (related or unrelated) person | 120 | 123 | 0 | 0 | 243
    Type of donor, Period 2: number analyzed (Participants) | 0 | 0 | 197 | 197 | 394
    Type of donor, Period 2: Donation after brain death | 0 | 0 | 66 | 65 | 131
    Type of donor, Period 2: Donation after circulatory death | 0 | 0 | 65 | 69 | 134
    Type of donor, Period 2: Donation from living (related or unrelated) person | 0 | 0 | 66 | 63 | 129
Donor sex [Count of Participants; unit: Participants] — Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Participants
    number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    Male | 215 | 207 | 0 | 0 | 422
    Female | 193 | 179 | 0 | 0 | 372
    Unknown | 18 | 40 | 0 | 0 | 58
Cold ischaemia time (h) [Mean (Standard Deviation); unit: Hours] — For deceased donor transplants only. Population: Period 1: Baseline data (852 participants) at randomization to induction therapy (Alemtuzumab or Basiliximab).
  Period 2: 6-months post-transplantation, baseline data (394 of the original participants) at re-randomization to maintanence therapy (Sirolimus or Tacrolimus).
  Hours
    number analyzed (Participants) | 426 | 426 | 0 | 0 | 852
    (all) | 13.9 (5.7) | 12.9 (6.0) |  |  | 13.4 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy-proven Acute Rejection at 6-months After Randomization to Induction Therapy
Description: Occurence of biopsy-proven acute rejection events at 6-months after transplantation during Period 1 (randomization to induction therapy (Campath-1H and Tacrolimus, or Basiliximab and Tacrolimus))
Time Frame: 6 months post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus
Number analyzed (Participants) | 426 | 426
Participants | 31 | 68
Statistical Analysis 1: Comparison: Period 1: Alemtuzumab/Tacrolimus vs Period 1: Basiliximab/Tacrolimus; Test type: Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.28 to 0.64]

2. Primary Outcome: Graft Function (at 18-months After Randomization to Maintenance Therapy)
Description: Estimated glomerular filtration rate (estimated using MDRD formula) at 18-months after maintenance therapy randomization to either Sirolimus or Tacrolimus.
Time Frame: 2 years post-transplantation
Measure: Mean (Standard Error); unit: mL/min/1.73m²
Arm/Group | Period 2: Sirolimus | Period 2: Tacrolimus
Number analyzed (Participants) | 197 | 197
mL/min/1.73m² | 53.7 (0.9) | 54.6 (0.9)
Statistical Analysis 1: Comparison: Period 2: Sirolimus vs Period 2: Tacrolimus; Test type: Other; p = 0.5, ANCOVA

3. Secondary Outcome: Number of Participants With Graft Failure (at 6-months After Randomization to Induction Therapy)
Description: Return to dialysis or re-transplantation by 6-months after randomization to induction therapy.
Time Frame: 6 months post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus
Number analyzed (Participants) | 426 | 426
Participants | 16 | 13
Statistical Analysis 1: Comparison: Period 1: Alemtuzumab/Tacrolimus vs Period 1: Basiliximab/Tacrolimus; Test type: Other; p = 0.58, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.59 to 2.55]

4. Secondary Outcome: Number of Participants With Graft Failure (at 18-Months After Randomization to Maintenance Therapy)
Description: Return to dialysis or re-transplantation by 18-months after randomization to maintenance therapy.
Time Frame: 2 years post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: Sirolimus | Period 2: Tacrolimus
Number analyzed (Participants) | 197 | 197
Participants | 8 | 4
Statistical Analysis 1: Comparison: Period 2: Sirolimus vs Period 2: Tacrolimus; Test type: Other; p = 0.23, Log Rank; Rate Ratio = 1.99, 95% CI 2-sided [0.64 to 6.18]

5. Secondary Outcome: Number of Participants With Serious Infection (at 6-months After Randomization to Induction Therapy)
Description: Occurrence of any serious infection (opportunistic or requiring admission to hospital) reported within Period 1 (randomization to induction therapy of either Alemtuzumab (Campath-1H) and Tacrolimus, or Basiliximab and Tacrolimus).
Time Frame: 6-months post-transplantation
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Campath 1H/Tacrolimus: Induction therapy allocation: Campath-1H and Tacrolimus
  Alemtuzumab: Alemtuzumab 30 mg intravenously or subcutaneously, two doses 24 hours apart
  Tacrolimus: Target trough level 5-7 ng/mL for 6-months after alemtuzumab.
Arm/Group | Period 1: Campath 1H/Tacrolimus | Period 1: Basiliximab/Tacrolimus
Number analyzed (Participants) | 426 | 426
Participants | 135 | 136
Statistical Analysis 1: Comparison: Period 1: Campath 1H/Tacrolimus vs Period 1: Basiliximab/Tacrolimus; Test type: Other; p = 0.88, Regression, Cox; Rate Ratio = 1.02, 95% CI 2-sided [0.80 to 1.29]

6. Secondary Outcome: Number of Participants With Serious Infection (at 18-months After Randomization to Maintenance Therapy)
Description: Occurrence of any serious infection (opportunistic or requiring admission to hospital) reported during Period 2 (maintenance therapy randomization to either Sirolimus or Tacrolimus).
Time Frame: 2 years post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: Sirolimus | Period 2: Tacrolimus
Number analyzed (Participants) | 197 | 197
Participants | 95 | 70
Statistical Analysis 1: Comparison: Period 2: Sirolimus vs Period 2: Tacrolimus; Test type: Other; p = 0.008, Log Rank; Rate ratio = 1.51, 95% CI 2-sided [1.11 to 2.06]

7. Secondary Outcome: Number of Participants With Cancer (at 18-months After Randomization to Maintenance Therapy)
Description: Occurrence of any cancer reported during Period 2 (maintenance therapy randomization to either Sirolimus or Tacrolimus).
Time Frame: 2 years post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: Sirolimus | Period 2: Tacrolimus
Number analyzed (Participants) | 197 | 197
Participants | 17 | 17
Statistical Analysis 1: Comparison: Period 2: Sirolimus vs Period 2: Tacrolimus; Test type: Other; p = 0.99, Log Rank; Rate Ratio = 1.00, 95% CI 2-sided [0.51 to 1.97]

8. Secondary Outcome: Number of Participants With Major Vascular Event (at 18-months After Randomization to Maintenance Therapy)
Description: Composite of non-fatal myocardial infarction, non-fatal stroke, cardiovascular death or arterial revascularization
Time Frame: 2 years post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: Sirolimus | Period 2: Tacrolimus
Number analyzed (Participants) | 197 | 197
Participants | 10 | 13
Statistical Analysis 1: Comparison: Period 2: Sirolimus vs Period 2: Tacrolimus; Test type: Other; p = 0.52, Log Rank; Rate Ratio = 0.76, 95% CI 2-sided [0.34 to 1.73]

ADVERSE EVENTS:
Time Frame: Period 1: SAEs collected during the 6-months post-transplantation Period 2: SAEs collected between 6-months and 24-months post-transplantation
Description: Information about the occurrence of serious adverse events was recorded at scheduled visits
  Other (not including Serious) Adverse Events were not recorded or assessed.
Groups:
- Period 2: Sirolimus: Maintenance therapy allocation: Sirolimus
  Target trough level of 6-12 ng/mL for the first 6-months then reducing to 5-10 ng/nL
- Period 2: Tacrolimus: Maintenancy therapy allocation: Tacrolimus
  Target trough level of 5-7 ng/mL
Arm/Group | Period 1: Alemtuzumab/Tacrolimus | Period 1: Basiliximab/Tacrolimus | Period 2: Sirolimus | Period 2: Tacrolimus
All-Cause Mortality (participants affected / at risk) | 11/426 | 6/426 | 11/197 | 9/197
Serious Adverse Events (participants affected / at risk) | 341/426 | 354/426 | 140/197 | 134/197
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Alemtuzumab/Tacrolimus (N=426) | Period 1: Basiliximab/Tacrolimus (N=426) | Period 2: Sirolimus (N=197) | Period 2: Tacrolimus (N=197)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 26 | 15 | 3 | 7
Cardiac disorders (Cardiac disorders) | 14 | 15 | 10 | 3
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Endocrine disorders (Endocrine disorders) | 0 | 0 | 0 | 0
Eye disorders (Eye disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 39 | 40 | 27 | 25
General disorders and administration site conditions (General disorders) | 22 | 13 | 5 | 2
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1 | 3 | 2
Immune system disorders (Immune system disorders) | 41 | 70 | 33 | 9
Infections and infestations (Infections and infestations) | 158 | 161 | 97 | 74
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 154 | 131 | 13 | 7
Investigations (Investigations) | 140 | 136 | 24 | 26
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 20 | 23 | 19 | 18
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 4
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 18 | 17
Nervous system disorders (Nervous system disorders) | 10 | 13 | 8 | 13
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0
Psychiatric disorders (Psychiatric disorders) | 5 | 2 | 0 | 1
Renal and urinary disorders (Renal and urinary disorders) | 24 | 37 | 7 | 9
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 | 15 | 7 | 4
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 4
Social circumstances (Social circumstances) | 0 | 0 | 0 | 0
Surgical and medical procedures (Surgical and medical procedures) | 190 | 190 | 39 | 35
Vascular disorders (Vascular disorders) | 13 | 14 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan: Induction Therapy Data Analysis Plan (2014-02-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT01120028/SAP_000.pdf
  • Study Protocol (2011-12-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT01120028/Prot_001.pdf
  • Statistical Analysis Plan: Maintenance Therapy Data Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT01120028/SAP_002.pdf